CLINICAL TRIAL: NCT04897386
Title: Monitoring the Efficacy of Duvalizumab Combined With Neoadjuvant Chemotherapy for Ib-IIIb NSCLC by Sequencing of Immune Receptor Repertoire: a Prospective, One Arm Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: duvalizumab
Record Dates: First submitted 2021-05-20; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Ib-IIIb NSCLC
MeSH Terms: interventions — Pemetrexed; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duvalizumab Combined With Neoadjuvant Chemotherapy (Experimental)
  Interventions: Drug: Duvalizumab

INTERVENTIONS:
Drug: Duvalizumab — Pemetrexed 850 mg, IV, Day1; Platinum 50mg / m2, IV, day1, once every 3 weeks, duvalizumab treatment, 1500mg, day1, a total of 4 cycles, once every 3 weeks. 4 cycles in total
  Other Names: Pemetrexed; platinum

SUMMARY:
To observe and evaluate the efficacy and safety of Duvalizumab Combined With Neoadjuvant Chemotherapy for Ib-IIIb NSCLC and the relevance with Immune Receptor Repertoire

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old;
2. NSCLC confirmed by histopathology;
3. According to the doctor's advice, according to the routine diagnosis and treatment process, lung cancer patients who need radical resection and neoadjuvant therapy before operation;
4. No previous treatment for esophageal cancer, including surgery, chemotherapy, radiotherapy, targeted therapy, hormone or immunotherapy;
5. ECoG score was 0 or 1;
6. There was no operative contraindication in preoperative organ function examination;
7. At least 6 months of expected survival
8. The laboratory examination met the following standards:

   1. Bone marrow function: hemoglobin (HB) ≥ 90g / L; White blood cell count (WBC) ≥ the lower limit of normal value; Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L； Platelet count ≥ 90 × 10^9/L；
   2. Renal function: Cr ≤ unl (upper limit of normal value) × 5, CCR ≥ 55ml / min;
   3. Liver function: total bilirubin ≤ ULN × 1.5； ALT and AST ≤ ULN × 2.5 (patients with liver metastasis can be relaxed to ≤ 5 * ULN);
   4. Coagulation function: international normalized ratio of prothrombin time ≤ ULN × 5, and partial thromboplastin time was within the normal range;
9. The subjects agreed and voluntarily signed the informed consent

Exclusion Criteria:

1. Allergic to the study drug;
2. History of hemorrhagic disease or with hemorrhagic disease
3. Liver and kidney dysfunction;
4. Patients with uncontrolled diseases (including but not limited to: active infection, symptomatic congestive heart failure; Myocardial infarction occurred within 3 months; Unstable angina, arrhythmia, etc.);
5. Women of childbearing age are unwilling to use contraception;
6. Lactating women;
7. For any other reason, the researchers consider it inappropriate to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | at 64th week
  Objective response rate
DFS | at 64th week
  disease free survival